CLINICAL TRIAL: NCT05420064
Title: Digital Technology to Enhance Access to and Effectiveness of Cancer Genetic Counseling: Effective Familial OutReach Via Tele-genetics (EfFORT) Trial & Supporting Test Result Interpretation and Variant Education (STRIVE) Trial
Brief Title: An Intervention to Increase Genetic Testing in Families Who May Share a Gene Mutation Related to Cancer Risk and An Intervention to Help Patients and Their Primary Care Providers Stay Up-to-date About Uncertain Genetic Test Results
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-023
Record Dates: First submitted 2022-06-06; First posted 2022-06-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: BRCA1 Mutation; POLD1 Gene Mutation; CDKN2A Mutation; BRCA2 Mutation; POLE Gene Mutation; APC Gene Mutation; ATM Gene Mutation; MLH1 Gene Mutation; BARD1 Gene Mutation; MSH2 Gene Mutation; BRIP1 Gene Mutation; MSH6 Gene Mutation; CHEK2 Gene Mutation; PMS2 Gene Mutation; PALB2 Gene Mutation; EPCAM Gene Mutation; RAD51C Gene Mutation; BMPR1A Gene Mutation; RAD51D Gene Mutation; SMAD4; PTEN Gene Mutation; GREM1
Keywords: EfFORT; Memorial Sloan Kettering Cancer Center; Genetic Testing; 22-023
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Proband-Mediated Cascade Genetic Testing (Active Comparator): Control arm- Behavioral: As per standard of care, probands will be given a Family Letter by their genetic counselor that they will be instructed to share with their at-risk relatives (ARR). In addition to the recommendation that ARR undergo genetic counseling and a list of local genetics clinics, this letter will include a link to the eDGP through which control ARR can enroll onto the present study. For these ARR, the eDGP will only be used to obtain study e-consent and to administer study surveys.
  Interventions: Behavioral: Standard of Care
- EfFORT Trial Intervention Arm: Provider-Facilitated Cascade Genetic Testing (Experimental): Intervention arm-: Behavioral: Probands will give contact info for their ARR in the eDGP and indicate a date by which they will discuss the familial pathogenic variant with their ARR (can request a delay/halt to outreach). After this date the team will contact the ARR to invite them to review education and e-consent to the study. The study team will facilitate ARR cascade testing through telegenetics pre- and post-test counseling and saliva-based at home testing through MSK or a reference laboratory.
  Interventions: Behavioral: Intervention Arm At-risk Relative/ARR Contacts
- STRIVE Trial Control Arm: Patient-Led VUS Follow-Up (Active Comparator): Patients will receive standard of care post-test genetic counseling and discussion of implications for relatives, if any. Consistent with standard practice, most patients will likely be recommended against telling their relatives to seek genetic testing for the Variant of uncertain significance/VUS because it is not clinically useful. All participants with a VUS will be recommended to re-contact the MSK CGS in 1-2 years for updated information related to the VUS result
  Interventions: Behavioral: Standard of Care
- STRIVE Trial Intervention Arm: Digitally-Facilitated VUS Follow-Up (Experimental): Following standard of care post-test genetic counseling, patients will be provided access to the MyGene Portal. Through this portal, participants will be able to continuously engage with interactive educational materials including information about Variant of uncertain significance/VUS results and recommendations, access tools for participants to communicate with the CGS team, access the interactive pedigree (FamGenix) to provide updates about personal/family medical history, receive notifications about VUS reclassification, and receive reminders to self-schedule a follow-up clinical visit to discuss updates. In this way, participants will have a transparent, ongoing, and structured follow-up plan for their VUS management.
  Interventions: Behavioral: MyGene Portal
- EfFORT Trial De-Identified Non-Randomized Control Arm (No Intervention): This control arm is comparable to true standard of care.

INTERVENTIONS:
Behavioral: Intervention Arm At-risk Relative/ARR Contacts — Probands will give contact info for their ARR in the eDGP and indicate a date by which they will discuss the familial pathogenic variant with their ARR (can request a delay/halt to outreach). After this date the team will contact the ARR to invite them to review education and e-consent to the study. The study team will facilitate ARR cascade testing through telegenetics pre- and post-test counseling and saliva-based at home testing through MSK or a reference laboratory.
  Arms: EfFORT Trial Intervention Arm: Provider-Facilitated Cascade Genetic Testing
Behavioral: MyGene Portal — Through the MyGene Portal, participants will be able to continually access their genetic test results, personalized medical management recommendations from the MSK CGS care team, an interactive pedigree for personal/family history updates, and tailored educational materials for patients with a VUS in an effort to promote sustained engagement and transparency.
  Arms: STRIVE Trial Intervention Arm: Digitally-Facilitated VUS Follow-Up
Behavioral: Standard of Care — Participants will received appropriate clinical care as outline by standard of care guidelines
  Arms: Proband-Mediated Cascade Genetic Testing; STRIVE Trial Control Arm: Patient-Led VUS Follow-Up

SUMMARY:
The purpose of this study is to examine the impact of new cancer genetic counseling models that aim to increase patient engagement with the genetics team. To do this, the study consists of two trials to evaluate two related interventions. The first trial is the EfFORT Trial, which evaluates a cascade genetic testing intervention. Cascade testing is the process of offering genetic testing to people who are at risk of having inherited a possibly harmful gene change that has been found in their family. The study will look at how often genetic testing occurs when healthcare providers have permission to reach out to family members to recommend genetic testing and to help those who are interested get tested. The study will look at whether this cascade testing intervention is practical and effective. The study would like to see how this approach of healthcare providers reaching out directly to family members compares with the usual approach of patients telling their family members about the recommendation to get genetic testing. The second trial is the STRIVE Trial, which evaluates an intervention designed to help patients who receive an uncertain result from genetic testing (also called a "variant of uncertain significance") stay connected with their genetics care team, and to help patients and their primary care providers stay up-to-date about the meaning of uncertain genetic test results. The study will look at whether an intervention that consists of a study online portal for patients with uncertain genetic test results and their primary care providers will help them to stay up-to-date on the meaning of uncertain genetic test results. The study would like to see how this intervention compares to the usual approach of encouraging patients to re-contact their genetics care team on their own about a year after getting genetic testing."

ELIGIBILITY:
Inclusion Criteria:

EfFORT Trial Probands

* Current MSK patient
* Received post-test genetic counseling from MSK Clinical Genetics Service within the last 3 months (or within the last year for the de-identified non-randomized control probands)
* 25 years of age or older
* Self-reported "very well" comprehension of written and verbal English language or Spanish language
* Has at least one ARR who meets criteria for study enrollment (see below)
* First in the family to test positive for PV at MSK in any of the following cancer susceptibility genes, or an ARR of an MSK proband who converted to the proband role:

APC I1307K, ATM, BARD1, BMPR1A, BRCA1, BRCA2, BRIP1, CDKN2A (P16), CHEK2, EPCAM, GREM1, MLH1, MSH2, MSH6, PALB2, PMS2, POLD1, POLE, PTEN, RAD51C, RAD51D, SMAD4, BAP1, DICER1, FH, FLCN, HOXB13, KIT, MAX, MEN1, MET, MITF, PTCH1, RAD51B, RET, SDHB, SDHC, SDHD, STK11, SUFU, TMEM127, TSC1, TSC2, VHL

Principal Investigator discretion will be used to determine whether specific variants within the above genes meet a clinical actionability threshold to warrant familial genetic testing.

EfFORT Trial At-Risk Relatives (ARRs):

* Biological first-, second-, or third- degree relative of enrolled MSK proband
* 25 years of age or older
* Resides within the United States
* Self-reported medical insurance which can be in or out of network with MSK
* Self-reported "very well" comprehension of written and verbal English language

STRIVE Trial VUS Patients

* Current MSK patient
* Received post-test genetic counseling from MSK Clinical Genetics Service within the last 3 months
* 25 years of age or older
* Self-reported "very well" comprehension of written and verbal English language or Spanish language
* Has a VUS identified in any of the following cancer predisposition genes:

APC, ATM, AXIN2, BAP1, BARD1, BLM, BMPR1A, BRCA1, BRCA2, BRIP1, CDH1, CDK4, CDKN2A (P16), CHEK2, CTNNA1, DICER1, ELOC, EPCAM, FH, FLCN, GREM1, HOXB13, KEAP1, MAX, MBD4, MEN1, MET, MITF, MLH1, MLH3, MSH2, MSH3, MSH6, MUTYH, NF1, NF2, NTHL1, PALB2, PMS2, POLD1, POLE, POT1, PTEN, RAD51B, RAD51C, RAD51D, RB1, RET, RNF43, RPS20, SDHA, SDHAF2, SDHB, SDHC, SDHD, SMAD4, STK11, TERT, TMEM127, TP53, TSC1, TSC2, VHL

STRIVE Trial PCP Providers:

* Designated healthcare provider for an enrolled VUS patient
* Resides within the United States

Exclusion Criteria:

EfFORT Trial Probands

* Is unwilling or unable to provide informed consent
* Is unwilling or unable to create a MyMSK patient portal account (see section 3.0 on MyMSK patient usage at MSK and CGS)
* Does not have an email address
* Has enrolled in the STRIVE trial

EfFORT Trial At-Risk Relatives (ARRs):

* Is unwilling or unable to provide informed consent
* Is unwilling or unable to create a MyMSK patient portal account
* Has previously undergone genetic testing for the familial PV
* Does not have an email address
* Has opted out of study contact

STRIVE Trial VUS Patients

* Is unwilling or unable to provide informed consent
* Is unwilling or unable to create a MyMSK patient portal account (see section 3.0 on MyMSK patient usage at MSK and CGS)
* Does not have an email address
* Has enrolled in the EfFORT trial

STRIVE Trial PCP Providers

* Contact information not available

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of genetic testing uptake in provider-facilitated cascade testing intervention to the proband-mediated cascade testing control | 12 months
  The Primary Objective for EfFORT Trial: Assess genetic testing uptake by first-, second-, and third-degree relatives in the provider-facilitated cascade testing intervention as compared to the proband-mediated cascade testing control.
Comparison of participant perceived quality of care | 12 months
  The Primary Objective for STRIVE Trial: Assess perceived quality of Variant of uncertain significance/VUS follow-up care and continued engagement with the Clinical Genetics Service/CGS care team in the digitally-facilitated VUS follow-up intervention as compared to the patient-led VUS follow-up control. A modified subset of items based upon an existing survey of patient-centered quality of follow-up care for cancer survivors (Cronbach's α=0.65-0.93) will be used to measure patient perceptions of the quality of their follow-up care provided by both the CGS care team (11 items) and their PCPs (6 items). Items are measured on a 4-point Likert-type scale, and mean scores are computed such that higher scores indicate greater perceived quality of care This measure will be collected from VUS patient participants in both study arms and a mean score calculated across items.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activity), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK at Ralph Lauren (Limited Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activity), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org